CLINICAL TRIAL: NCT03143374
Title: Positron Emission Tomography (PET) Imaging of Tau Pathology in Neurodegenerative Disease
Brief Title: PET Tau - Neurodegenerative Disease Imaging
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 824867
Record Dates: First submitted 2016-11-02; First posted 2017-05-08 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Neurodegenerative Disease
Keywords: Neurodegenerative Disease
MeSH Terms: conditions — Neurodegenerative Diseases | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Positron Emission Tomography (PET/CT) Imaging of Tau Pathology in Neurodegenerative Disease (Experimental): Individuals who have been diagnosed with FTD, PPA, CBD, PSP, MCI, AD, PCA, PD, PDD, DLB, MSA, ALS or FTD-ALS may participate in this study if they are 18 years of age or older; most participants will be receiving care at the clinical practices of the of the University of Pennsylvania and at Pennsylvania Hospital Department of Neurology. Healthy control subjects will also be recruited for this study.
  Interventions: Drug: 18F-AV-1451

INTERVENTIONS:
Drug: 18F-AV-1451 — The experimental tracer used for this study is called 18F-AV-1451 is a specialized radioactive PET tracer used to detect the presence of tau proteins in the brain.
  Participants will undergo a baseline 18F-AV-1451 brain scan. If funding is available, participants will be asked to return for one or more longitudinal visits, including a 18F-AV-1451 brain scan, every 9 to 18 months after the prior visit.
  The 18F-AV-1451 PET/CT scan will require up to 3 hours of time, including preparation. The scan will take place using PET/CT scanners in the Perelman Center for Advanced Medicine or the Hospital of the University of Pennsylvania.
  Other Names: formally known as 18F-T807; 7-(6-[18F]fluoropyridin-3-yl)-5H-pyrido[4,3-b]indole

SUMMARY:
The purpose of this study is to measure the amount of a protein in the brain known as tau using an imaging procedure called Positron Emission Tomography (PET/CT). Tau has been shown to build up in the brains of patients with injury to brain cells. This study looks at neurodegenerative diseases such as frontotemporal degeneration (FTD).

DETAILED DESCRIPTION:
The purpose of this study is to measure the amount of a protein in the brain known as tau using an imaging procedure called Positron Emission Tomography (PET/CT). Tau has been shown to build up in the brains of patients with injury to brain cells, including Alzheimer's disease, Parkinson's disease, Lewy body disease and Frontotemporal degeneration. 18F-AV-1451 (formally known as 18F-T807) is a specialized radioactive PET tracer that sticks to the tau protein in the brain. In this study, researchers will use 18F-AV-1451 to form images of tau binding in the brain. 18F-AV-1451 is an investigational or experimental imaging agent that has not yet been approved by the Food and Drug Administration for use in brain imaging.

In this study, researchers want to find out how accurate and useful 18F-AV-1451 is in imaging patients who have problems with thinking, remembering, speech, and visual activities, and may be diagnosed with different types of neurodegenerative disease. This study will help test how imaging measures may provide information that could be used to determine diagnosis for patients in the future. The results of the PET/CT scan will be compared with other information obtained under related protocols, including brain magnetic resonance imaging (MRI), spinal fluid and cognitive test results.

ELIGIBILITY:
INCLUSION CRITERIA FOR NEURODEGENERATIVE SUBJECTS

1. Participants has been diagnosed with one of the following neurodegenerative diseases: FTD, PPA, CBD, PSP, MCI, AD, PCA, PD, PDD, DLB, MSA, ALS or FTD- ALS
2. Participants will be 18 years of age or older
3. Participants must be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study-specific procedures. If the subject is unable to provide informed consent, the subject's legal representative may consent on behalf of the patient, but the patient will be asked to confirm assent.
4. Participants must be willing and able to comply with scheduled visits and imaging procedures.
5. Subject is concurrently enrolled in centers UNICORN(842873) protocol.

INCLUSION CRITERIA FOR HEALTHY CONTROL SUBJECTS

1. Participants will be 18 years of age or older.
2. Participants must be informed of the investigational nature of this study and provide written informed consent in accordance with institutional and federal guidelines prior to study-specific procedures.
3. Participants must be willing and able to comply with scheduled visits and imaging procedures.
4. Subject is concurrently enrolled in centers UNICORN(842873) protocol

EXCLUSION CRITERIA FOR ALL SUBJECTS

1. Females who are pregnant or breast feeding at the time of the baseline PET/CT scan will not be eligible for this study. A urine pregnancy test will be performed in women of child-bearing potential at screening and within 24 hours of any scheduled PET/CT.
2. Inability to tolerate or contraindication to imaging procedures in the opinion of an investigator or treating physician
3. Any medical or psychological condition that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study
4. The investigators may choose to exclude participants with clinically significant cardiovascular disease and/or documented abnormalities on ECG out of an abundance of caution.
5. The investigators of UNICORN (IRB #842873) have determined the participant has evidence of structural abnormalities such as major stroke or mass on MRI that is likely to interfere with analysis of the PET scan.

ADDITIONAL EXCLUSION CRITERIA FOR HEALTHY CONTROL SUBJECTS

1. Pre-existing psychiatric conditions (e.g., active depression, schizophrenia, or active anxiety) or neurological conditions (e.g., stroke, epilepsy, head trauma) per medical record review or self-report.
2. Current use of psychoactive medications or substances per medical record review or self-report.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-08-23 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Regional uptake | 10 years
  Examine regional anatomic distribution of PET-tau uptake comparatively in dementia syndromes and PET-Tau uptake with neuropsychology and MRI regional GM atrophy at baseline collected under other center protocols. Uptake with neuropsychology and MRI regional GM atrophy at baseline.

SECONDARY OUTCOMES:
Changes over time | 10 years
  Use regression to relate longitudinal neuropsychological and regional MRI decline in dementia syndromes to baseline regional PET-tau uptake.
CSF Correlate | 10 years
  Correlate CSF total and phosphorylated (p-tau/t-tau) tau with regional PET-tau uptake in dementia syndromes at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: David Irwin, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No